CLINICAL TRIAL: NCT01792908
Title: Has Kinesio Tape Effects on Ankle Proprioception? A Randomized Clinical Trial
Brief Title: Kinesio Tape Effects on Ankle Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Iris Miralles Rull, Lecturer, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T11230S; R02/2010 (Other Grant/Funding Number: Col.legi de Fisioterapeutes de Catalunya)
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Sprains and Strains
Keywords: ankle lateral ligament; athletic tape; position sense; Proprioception
MeSH Terms: conditions — Sprains and Strains | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KT group (Experimental): The KT group received ankle KT on the lateral ligament in the non-dominant leg and a recommendation guide. The Kinesio tape procedure was carried out by the same certified athletic therapist to ensure consistency throughout the study.
  Interventions: Device: Kinesio tape
- Control group (No Intervention): Any intervention has been applied. Using another kind of tape or a different KT application for control group may increase cutaneous information, undermining our goal.

INTERVENTIONS:
Device: Kinesio tape — The KT used was Kinesiology Tape® of 5 cm and it was applied according to Kase protocol (Kase K). The first layer of tape consisted of a single strip placed over the anterior talofibular ligament from insertion to origin, with a 50% tension, except the two-centimetre proximal and distal ends, applied with no tension. The same procedure was repeated for the calcaneofibular ligament and posterior talofibular ligament
  Other Names: Kinesio-tape; Kinesiotape; KinesioTM tape
  Arms: KT group

SUMMARY:
The aim of the present study was to establish whether Kinesio Tape (KT) on the ankle (Kase protocol for the lateral ankle ligament) improves Joint Position Sense (JPS) in healthy volunteers immediately after its application and 48 hours later.

DETAILED DESCRIPTION:
The investigators assessed Joint Position Sense (JPS) through the difference of error (DoE) and the deviation of the target angle (DTA). JPS was assessed before the Kinesio Tape (KT) was placed, immediately after and 48 hours later.

ELIGIBILITY:
Inclusion Criteria:

* Must be signed the informed consent
* Aged between 18 and 35 years
* Did not suffered from ankle or foot skin diseases
* Active dorsal/plantarflexion ARoM equal to or above 15º and inversion/eversion
* ARoM equal to or above 5º.

Exclusion Criteria:

* Traumatic, neurological or circulatory diseases diagnosed
* Joint laxity
* More than three ankle sprains in their lives or one in the last 12 months that required treatment and ankle or foot pain at the time of study enrolment in the non-dominant lower limb.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Joint position sense on the Difference of Error from the target angle | Change from baseline in proprioception at 48h
  The primary outcome, difference of error (DE) in degrees was calculated to show changes in error from the target angle over time. We compared error, before and immediately after intervention (DoE 1-2), before and 48 hours after intervention (DE 1-3) and immediately and 48 hours after intervention (DE 2-3).

SECONDARY OUTCOMES:
Deviation of the target angle | Change from baseline in proprioception at 48h
  We also calculated the deviation from the target angle (DTA) in degrees, this secondary outcome to describe the direction of error when subjects tried to reproduce the requested position. Deviation was obtained encoding net error taking as correct position when the target and the estimated angle were equal, considering the precision of the electronic plate a valid range (0.4 degrees). Values above this range were classified as Overestimation and as Underestimation when values were below this range.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Miralles, Principal Investigator — University Rovira i Virgili
Locations (1):
- Faculty of Medicina i Ciències de la Salut; University Rovira i Virgili., Reus, Tarragona, Spain

REFERENCES:
- [Background] Miralles I, Monterde S, Montull S, Salvat I, Fernandez-Ballart J, Beceiro J. Ankle taping can improve proprioception in healthy volunteers. Foot Ankle Int. 2010 Dec;31(12):1099-106. doi: 10.3113/FAI.2010.1099. PMID 21189212